CLINICAL TRIAL: NCT07182149
Title: A Phase 1a/1b Study of NRM-823 as Monotherapy and in Combination With Immune Checkpoint Inhibition in Participants With Locally Advanced or Metastatic Refractory Solid Tumors
Brief Title: A Phase 1 Study of NRM-823 in Participants With Locally Advanced or Metastatic Refractory Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Normunity AccelCo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRM-823-101
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: HNSCC; ESCC; Esophageal Adenocarcinoma; Gastric Adenocarcinoma; GEJ Adenocarcinoma; Ovarian Cancer; NSCLC; Cervical Cancer; Endometrial Cancer; Triple Negative Breast Cancer (TNBC)
Keywords: NRM-823
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Adenocarcinoma Of Esophagus; Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NRM-823 (Experimental): Administered per protocol requirements
  Interventions: Drug: NRM-823

INTERVENTIONS:
Drug: NRM-823 — NRM-823 is a bispecific T-Cell Engager

SUMMARY:
This study is being done to find out of NRM-823 is safe and can treat participants with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Part A of the study will evaluate the safety and tolerability of NRM-823. Part B of the study will further evaluate the safety and tolerability of NRM-823 of the recommended dose identified in PART A in an expansion cohort. Part C will evaluate the addition of a checkpoint inhibitor to NRM-823.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically- or cytologically-diagnosed NSCLC (squamous or adenocarcinoma), TNBC, HNSCC, ESCC, esophageal adenocarcinoma, gastric/GEJ adenocarcinoma, cervical, endometrial, or ovarian cancer which is advanced or metastatic.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Adequate liver, renal, pulmonary, and cardiac function.
* Adequate hematologic function.

Exclusion Criteria:

* Has received cytotoxic chemotherapy, biologic anticancer agents, checkpoint inhibitors, or radiation therapy (excluding bone-only radiation therapy) ≤3 weeks or 5 half-lives (whichever is shorter) prior to the first dose of NRM-823
* History of Grade 2 pneumonitis requiring steroids or any Grade 3 or 4 pneumonitis from any prior therapy.
* Has received an investigational therapy <4 weeks or 5 half-lives prior to the first dose of NRM823, whichever is shorter prior to the first dose of NRM-823.
* With the exception of alopecia and Grade ≤2 neuropathy, any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAE) | From enrollment until 30 days post the last dose received by a participant
  Number of participants who experience treatment emergent AEs or SAEs
Incidence of dose-limiting toxicities (DLTs) | From enrollment until 30 days post the last dose received by a participant
  Number of participants who experience a DLT. A DLTs include protocol defined adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Bozon, MD, Study Director — Normunity AccelCo, Inc.
Locations (9):
- United States (9):
  - Normunity Investigational Site, Denver, Colorado
  - Normunity Investigational Site, New Haven, Connecticut
  - Normunity Investigational Site, Minneapolis, Minnesota
  - Normunity Investigational Site, Maumee, Ohio
  - Normunity Investigational Site, Philadelphia, Pennsylvania
  - Normunity Investigational Site, Nashville, Tennessee
  - Normunity Investigational Site, Dallas, Texas
  - Normunity Investigational Site, San Antonio, Texas
  - Normunity Investigational Site, Fairfax, Virginia